CLINICAL TRIAL: NCT02985931
Title: Single-scan Rest/Stress Imaging With Cadmium Zinc Telluride-based SPECT for Coronary Flow Quantification
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tzu-Chen Yen, Professor, Chang Gung Memorial Hospital
Other Study IDs: 101-0453A3
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Quantitative Analysis of SPECT MPI
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected CAD subjects
  Interventions: Other: Diagnostic imaging scans of SPECT and MRI

INTERVENTIONS:
Other: Diagnostic imaging scans of SPECT and MRI

SUMMARY:
The investigators aim to address this issue with novel image quantification methods using CZT-based SPECT, which is capable of dynamic data acquisition and therefore feasible for the quantification of the coronary flow. The investigators will use kinetic modeling techniques to design a study that allows the absolute flow quantification. To make this study practical, the investigators will develop a protocol that includes the acquisition of both the rest and stress scan within the same scan that is shorter than 30 minutes. The SPECT-measured flow will be validated against the flow measured with cardiac MRI scans. Patients with high CAD risk will be recruited for the clinical trial. Data from these human subjects will be used for determination of the performance of the developed algorithm. With the proposed rapid scan with absolute quantification capabilities, the investigators expect to increase the diagnosis accuracy while maintaining the patient throughput.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with high possibility of coronary artery disease after being evaluated by a cardiologist.
2. > 20 years old.
3. Not under infection or other conditions inappropriate for being recruited.
4. Without myocardial infarction within one week.
5. With stable blood pressure.
6. Subjects with normal kidney functions and without allergic reactions to MRI contrast agents.

Exclusion Criteria:

1. Subjects who cannot take a SPECT scan or do not agree to sign the informed consent.
2. Pregnant subjects or subjects who are currently breast-feeding.
3. Those currently under radiation therapies.
4. Patients with pleural effusion.
5. Patients who are allergic to SPECT tracers.
6. Patients with serious psychological disorders.
7. Patients with asthma.
8. Patients with stroke within a week.
9. Patients with AV block.
10. Patients with sinus syndrome.
11. Subjects who are currently under other clinical trials.
12. Subjects with poor kidney functions who are inappropriate for MRI contrast agents.
13. Subjects with pacemakers.
14. Subjects with Claustrophobia.
15. Subjects who cannot hold breath for cardiac MRI studies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are suspected with coronary artery diseases and need imaging exams.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Correlation between SPECT- and MRI-measured flow values | through study completion, an average of 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Chen Yen, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital